CLINICAL TRIAL: NCT06264869
Title: A Novel Approach of Interdental Guided Creeping Technique (IGCT) for Augmentation of Deficient Interdental Papillae: Randomized Clinical Trial
Brief Title: Interdental Guided Creeping Technique
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Ahmed Y Gamal, Professor of Oral Medicine, Periodontology and Oral Diagnosis, Faculty of Dentistry, Ain Shams University. Professor of Periodontology, College of Oral and Dental Surgery, Misr University for Science and Technology., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 141123
Record Dates: First submitted 2024-02-08; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Interdental Papilla Recession
Keywords: Interdental papilla loss; Interdental papilla deficiency; Interdental papilla recession; Black triangle; Connective tissue graft; Collagen membrane; Minimally Invasive Surgery; Tunneling Techniques; Creeping Attachment; Plastic periodontal surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IGCT + CTG (Experimental): Interdental guided creeping technique (IGCT) + Connective tissue graft (CTG)
  Interventions: Procedure: Interdental guided creeping technique (IGCT) and connective tissue graft (CTG)
- IGCT + CM (Experimental): Interdental guided creeping technique (IGCT) + Collagen membrane (CM)
  Interventions: Procedure: Interdental guided creeping technique (IGCT) and collagen membrane (CM)

INTERVENTIONS:
Procedure: Interdental guided creeping technique (IGCT) and connective tissue graft (CTG) — Interdental guided creeping technique (IGCT) and connective tissue graft (CTG)
  Arms: IGCT + CTG
Procedure: Interdental guided creeping technique (IGCT) and collagen membrane (CM) — Interdental guided creeping technique (IGCT) and collagen membrane (CM)
  Arms: IGCT + CM

SUMMARY:
The aim of this randomized clinical trial is to treat interdental papillary deficiency with minimally invasive interdental guided creeping technique (IGCT) comparing collagen membrane versus connective tissue graft.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients having interdental papilla deficiency.
* Good Oral Hygiene.
* Age range: 18 - 50 years.

Exclusion Criteria:

* Pregnancy or lactation.
* Smokers.
* Alcoholic patients and drug abusers.
* Handicapped and prisoners.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Black triangle height | Baseline, 1, 3 and 6 months.
  In mm

SECONDARY OUTCOMES:
Percentage of interdental papillary fill | Baseline, 1, 3 and 6 months.
  In %
Papillary gain, black triangle reduction | Baseline, 1, 3 and 6 months.
  In mm, %
Papillary height, attached gingiva width | Baseline, 1, 3 and 6 months.
  In mm
Pocket depth, clinical attachment level, keratinized tissue thickness | Baseline, 3 and 6 months.
  In mm
Plaque index | Baseline, 1, 3 and 6 months.
  Scores
Gingival index | Baseline, 1, 3 and 6 months.
  Scores
Duration of surgery | At time of surgery
  In minutes
Patient Reported Outcome | At the day of surgery and the 1st 10 days postoperative.
  VAS score for pain
Patient Reported Outcome | 1, 3 and 6 months.
  Patient satisfaction (score)

CONTACTS AND LOCATIONS:
Overall Officials: Ghada G A.GamalElDin, Dr., Principal Investigator — PhD Student of Periodontology, Faculty of Dentistry, Cairo University; Mohamed S. Morgan, Dr., Principal Investigator — Master Student of Periodontology, Faculty of Dentistry, Ain Shams University; Ahmed Y Gamal, Prof., Study Director — Professor of Oral Medicine, Periodontology and Oral Diagnosis - Faculty of Dentistry - Ain Shams University, Professor of Periodontology - College of Oral and Dental Surgery - Misr University for Science and Technology